CLINICAL TRIAL: NCT03471598
Title: Reliability, Validity and Responsiveness of the Upright Motor Control Test in Patients With Stroke
Status: Terminated | Type: Observational
Why Stopped: The COVID-19 pandemic held the candidates and/or participants back to join. The investigators also stopped recruiting for safety concern.
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, Bo-Jhen Chen, Physical Therapist, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: 06-XD13-045
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Impaired motor function is common after stroke. Individuals with stroke often exhibit synergic pattern that disturb daily function. It is crucial to identify the movement impairment in the clinical settings. Upright Motor Control Test (UMCT) is one of the tests developed to assess the selective movement control and functional strength in people with central nervous disorders. It can be used to reflect the impairment of motor function and evaluate changes of performance after treatment. Yet is little to know the clinimetrics of the UMCT on clinical utility. To date, only few researches explore that UMCT has some construct and criterion validity.

Therefore, this study aims to 1) establish the inter-rater reliability to administer the UMCT. 2) explore the correlation between the Fugl-Meyer Assessment of Motor Recovery after Stroke (FMA) and UMCT. 3). investigate whether the UMCT is able to predict the walking ability in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* First-ever, unilateral cerebral stroke within one month
* Being able to maintain standing for more than 10 seconds

Exclusion Criteria:

* Could not follow commands
* Deformity or fracture of lower limb
* Less than 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with first-ever, unilateral cerebral stroke within one month
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Upright Motor Control Test | 1 month
  6-18; higher score means better isolated joint control.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment of Motor Recovery after Stroke | 1 month
  UE scale:0-66; LE scale:0-34; higher score means better motor function.

OTHER OUTCOMES:
10 Meter Walk Test | 1, 3, 6, and 12 month
  Test the time required to complete 10 meters of walking.
6-Minutes-Waking-Test | 1, 3, 6, and 12 month
  Record the distance in six-minute walking.
Berg Balance Scale | 1, 3, 6, and 12 month
  score: 0-56; lower score means higher risk of fall.
Stroke Rehabilitation Assessment of Movement Measure | 1, 3, 6, and 12 month
  UE: 0-20; LE: 0-20: Mobility: 0-30; higher score indicated better motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Jhen Chen, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No